CLINICAL TRIAL: NCT02963844
Title: The Inspiratory Muscle Training Improves the Severity of Obstructive Sleep Apnea and Sleep Quality?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, José Carlos Nogueira Nóbrega Júnior, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08079697450
Record Dates: First submitted 2016-09-22; First posted 2016-11-15 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training (Experimental): The components of this group held the IMT load equivalent to 75% of the Pimáx. (measured weekly) for eight weeks.
  Interventions: Other: Inspiratory Muscle Training
- Inspiratory Muscle Training Sham (Sham Comparator): This group simulate the training, conducted the training without charge for the same period the intervention group.
  Interventions: Other: Inspiratory Muscle Training Sham

INTERVENTIONS:
Other: Inspiratory Muscle Training
  Other Names: Obstructive Sleep Apnea; Respiratory Muscle Training; Powerbreath
  Arms: Inspiratory Muscle Training
Other: Inspiratory Muscle Training Sham
  Other Names: No treatment
  Arms: Inspiratory Muscle Training Sham

SUMMARY:
Introduction: Obstructive sleep apnea (OSA) is characterized as a disorder that causes recurrent episodes of partial or complete obstruction of the upper airways during sleep. Objectives: In this way, the study will investigate the efficacy of inspiratory muscle training in improving the severity of obstructive sleep apnea and sleep quality of the research participants. Methods: The investigators will invite individuals of both sexes diagnosed with obstructive sleep apnea moderate and / or severe, arising from the Sleep Laboratory of the Hospital PROCAPE, located in Recife. This is a randomized-controlled trial, double-blind to be held in two groups: A) Individuals with OSA (moderate or severe) - Experimental Group: The components of this group hold the IMT with load of 75% of Pimáx. ( assessed weekly) for eight weeks. B) Individuals with OSA (moderate or severe) -Group control: This group will simulate training, performing no-load training for the same period the intervention group. All guidance on training and weekly evaluations will be made by the responsible for the research physiotherapist in Cardiopulmonary Physiotherapy Laboratory (LACAP - UFPE). Before and after the eight weeks, the groups will be evaluated by polysomnography, acoustic pharyngometry, tests for respiratory muscle strength (Manovacuometry) and lung function (spirometry). Expected results: Improvement of severity of OSA and sleep quality of research subjects after the completion of eight weeks of TMI when compared to the control group.

DETAILED DESCRIPTION:
Initially, the medical records of patients already submitted to PSG will be analyzed. Those classified as having moderate (15>AHI<30events/h) and severe (AHI>30events/h) OSA will be contacted by telephone to explain the procedure for participating in the research. Individuals who accept to participate in the study will be invited to attend the Cardiopulmonary Physiotherapy Laboratory and will perform an assessment consisting of collecting personal information through the application of a form, filling in the IPAQ and collecting anthropometric and vital signs data.

All members will be submitted to a polysomnography exam before and after the 8 weeks of training, in order to detect if there was a change in the AHI due to the training. The examination must be performed by the same physician responsible for interpreting the results and the diagnostic opinion, be conducted throughout the night, in spontaneous sleep, without any sedation or sleep deprivation. A computerized polysomnography system will be used to perform the exam. The parameters measured will be electrocardiogram (ECG), blood pressure (BP), chest and abdominal movements (plethysmography), peripheral oxygen saturation (SpO2) (pulse oximetry), nasal/buccal airflow (thermistors), body position and snoring ( MIC). In addition, the number of apneas, hypopneas, AHI and SpO2 levels will be calculated. The monitoring of pleasure or displeasure during the IMT session will be performed by applying the affective valence scale (AV), proposed by Hardy and Rejeski (1989). The scale is quantified from +5 to -5, corresponding, respectively, to the two antagonistic descriptors of the feeling during physical activity: "very good" and "very bad". In addition to these, the VA scale has intermediate descriptors: +3 = good; +1 = reasonably good; 0 = neutral; -1 = reasonably bad; -3 = bad. The scale will be answered by the volunteers at each weekly session performed with the physical therapist Subjects will complete the ESE before and after the 8 weeks of TMI. It is a scale containing eight daily situations requesting a self-assessment of the individual about the chance of dozing in the execution of these activities, scoring from 0 to 3, where 0: no chance of dozing, 1: small chance, 2: moderate chance, 3: high chance (ANNEX 2) (BERTOLAZI, ALESSANDRA NAIMAIER et al., 2009).

Subjects will complete the PSQI before and after the 8 weeks of TMI. It consists of a self-assessment questionnaire, which investigates sleep quality and disturbances over a period of 1 month. It consists of nineteen individual items that give rise to seven scoring "components": subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The sum of the scores obtained in the seven components generate a global score (BERTOLAZI, ALESSANDRA NAMAIER; BARRETO, 2008). Subjects will complete the SF-36 before and after the 8 weeks of IMT. It consists of a generic instrument for assessing quality of life, easy to administer and understand, but not as extensive as the previous ones. It is a multidimensional questionnaire formed by 36 items, encompassed in 8 scales or components: functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects, and mental health. It presents a final score from 0 to 100, in which 0 corresponds to the worst general health status and 100 to the best health status (ANNEX 4) (CICONELLI, 1999).

Subjects will complete the IPAQ prior to the TMI in order to assess their level of physical activity and ensure that only subjects classified as sedentary or insufficiently active are participating in the study. It is a questionnaire that makes it possible to estimate the time spent during the week with physical activities with moderate and strong intensity, in different contexts of daily life, such as: transport, work, performing household chores and leisure, as well as the time spent in passive activities, performed in the sitting position. The short version of the IPAQ contains seven open questions and its information allows estimating the time spent weekly in different spectra of physical activity (walking and physical efforts with moderate and strong intensities) and not performing physical activity (sitting position) (BERTOLDO BENEDETTI et al., 2007; MATSUDO et al., 2012). Subjects will perform manovacuometry before and weekly until completing 8 weeks of IMT. The present study will follow the recommendations proposed by the Thoracic Society/European Respiratory Society (ATS/ERS) and the Brazilian Society of Pneumology and Tisiology (SBPC), thus, during the collection of values referring to MIP and MEP, the patient will be seated, with the free arms and will be guided by the person responsible for carrying out the test to attach a mouthpiece (divers type) with a leak hole of 2mm of internal diameter to their mouth, the individual will be instructed to maintain an inspiratory and expiratory pressure for at least 1.5s in order to observe the maximum sustained pressure for one second (maximum mean pressure) in the manovacuometer (MVD 300, Globalmed, Brazil), used in the Cardiopulmonary Laboratory of the Department of Physiotherapy of the Federal University of Pernambuco (NEDER et al., 1999; ATS /ERS, 2002).

The test will be performed by an experienced operator who verbally encourages the subject to perform a maximal inspiratory effort against an occluded airway (Mueller maneuver) and a maximal expiratory effort against an occluded airway (Valsalva maneuver) at or near the residual volume ( RV) and total lung capacity (TLC respectively). The patient will be encouraged to perform the maneuvers to prevent air from escaping around the mouth, and will be instructed to hold the cheeks, if necessary, with the hands during the expiratory effort, as well as to press the lips firmly on the mouthpiece.

The three tests will be used (regardless of the order), which meet all the criteria considered acceptable. The measures with the highest value presented will be used (with variation less than or equal to 10% among the others). When the MIP values are identical, the one with the highest PPpeak value will be recorded, and successively the highest PPlatô and the lowest VPlatô

Some pulmonary function items will be evaluated before and weekly until completing the 8 weeks of IMT, described below:

* Slow vital capacity (SVC): it is measured during the expiration phase from the total lung capacity (TLC) or during inspiration from the residual volume (RV).
* Forced Vital Capacity (FVC): the patient will be asked to exhale as quickly and intensely as possible in a volume or flow spirometer after inhaling to full lung capacity. The exhaled volume can be read through the volume-time plot produced on a graph or derived from the flow integration. • Forced expiratory volume in one second (FEV1):
* Subsequently, the FEV1/VC and FEV1/FVC ratios will be calculated. The Berlin Questionnaire is considered as one of the most used tools to assist in OSA screening. The Berlin questionnaire in April 1996 and validated by Netzer et al in 1999. It is composed of self-administered questions, divided into three categories. Category 1 refers to the presence of snoring, category 2 assesses daytime sleepiness and falling asleep during daily activities, and category 3 looks at the history of Systemic Arterial Hypertension (SAH) and calculates the Body Mass Index (BMI) ( NETZER; STOOHS; NETZER, et al., 1999) After the initial assessment, patients will follow an intervention protocol for eight weeks using powerbreathe® (classic Light Resistance), a device capable of providing linear resistance in the inspiratory phase. . In the learning session (1st contact), the variables heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be monitored in order to provide greater safety during exercise and the physical therapist will guide how to perform of the exercise and the other sessions will be carried out by the individual at his/her home.

Subjects in both groups (intervention and placebo) will perform the training seated, using a nose clip, performing three cycles of thirty incursions, twice a day, seven days a week. For the intervention group set at 40% of MIP. and load ≤10% of MIP will be maintained. for individuals in the placebo group (value considered lower than the baseline level so that there is, in fact, training).

Another evaluator will adjust the load intensity weekly by evaluating MIP throughout the intervention protocol stage, so that blinding is preserved (CHARUSUSIN et al., 2013).

After the randomization process is carried out using the random allocation software, the individuals will receive a training diary from the researcher, to record the time of the exercises, the possible discomforts or difficulties of realization that may happen and for there to be a control of the execution of the training.

Each patient will receive a device (powerbreathe®) to carry out the training and the necessary guidelines for the training to take place at home. The necessary adjustments for the applied load will be made by the researcher through weekly meetings, respecting the individual needs of each patient, which will be determined by the advancement or not of the effort tolerance.

The first phase of the research will begin after the signing of the Free and Informed Consent Term (ICF), the physical evaluation and submission to the other tests, where each patient will be evaluated and guided to perform the proposed exercises that will be determined according to the ability of each individual.

The two groups will perform the training twice a day, however, the individuals in the control group will only use load <10% of their PI max and the intervention group will be subjected to a load of 40% of their PI max value.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with OSA (moderate or severe) by polysomnography;
* Be aged between 30 and 65;
* Sedentary or insufficiently active according to the International Physical Activity Questionnaire (IPAQ);
* Who are able to complete the proposed protocol;
* Individuals with BMI ≥ 18 ≤ 39.9 kg / m2.

Exclusion Criteria:

* Patients in non-invasive ventilation use (NIV);
* Individuals with account of orthopedic problems, neurological or cardiovascular or respiratory disease in your medical history that may cause obstruction during the stages of the research;
* Patients with BMI> 40 kg / m2.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2020-11 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Polysomnography - Apnea Hypopnea Index | 8 weeks
  number of apneas and hypopneas

SECONDARY OUTCOMES:
Sleep quality index of Pittsburgh - Sleep Quality | 8 weeks
  sleep quality grade

CONTACTS AND LOCATIONS:
Overall Officials: JOSE CARLOS NN JUNIOR, M.D., Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Per, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sengul YS, Ozalevli S, Oztura I, Itil O, Baklan B. The effect of exercise on obstructive sleep apnea: a randomized and controlled trial. Sleep Breath. 2011 Jan;15(1):49-56. doi: 10.1007/s11325-009-0311-1. Epub 2009 Nov 7. PMID 19898884
- [Background] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. The effect of exercise training on obstructive sleep apnea and sleep quality: a randomized controlled trial. Sleep. 2011 Dec 1;34(12):1631-40. doi: 10.5665/sleep.1422. PMID 22131599
- [Background] Charususin N, Gosselink R, Decramer M, McConnell A, Saey D, Maltais F, Derom E, Vermeersch S, van Helvoort H, Heijdra Y, Klaassen M, Glockl R, Kenn K, Langer D. Inspiratory muscle training protocol for patients with chronic obstructive pulmonary disease (IMTCO study): a multicentre randomised controlled trial. BMJ Open. 2013 Aug 5;3(8):e003101. doi: 10.1136/bmjopen-2013-003101. PMID 23921069
- [Background] Carneiro G, Florio RT, Zanella MT, Pradella-Hallinan M, Ribeiro-Filho FF, Tufik S, Togeiro SM. Is mandatory screening for obstructive sleep apnea with polysomnography in all severely obese patients indicated? Sleep Breath. 2012 Mar;16(1):163-8. doi: 10.1007/s11325-010-0468-7. Epub 2011 May 29. PMID 21626286
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Chien MY, Wu YT, Lee PL, Chang YJ, Yang PC. Inspiratory muscle dysfunction in patients with severe obstructive sleep apnoea. Eur Respir J. 2010 Feb;35(2):373-80. doi: 10.1183/09031936.00190208. Epub 2009 Jul 30. PMID 19643936
- [Result] Vranish JR, Bailey EF. Inspiratory Muscle Training Improves Sleep and Mitigates Cardiovascular Dysfunction in Obstructive Sleep Apnea. Sleep. 2016 Jun 1;39(6):1179-85. doi: 10.5665/sleep.5826. PMID 27091540